CLINICAL TRIAL: NCT04627766
Title: Validation of Continuous Monitoring of Vital Signs in Children With VTPatch Connected Device in the Pediatric Intensive Care Unit
Brief Title: Validation of Continuous Monitoring of Vital Signs in Children With a Connected Patch
Acronym: VITALPICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Philippe Jouvet, Professor, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-3157
Record Dates: First submitted 2020-11-09; First posted 2020-11-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Vital Signs
Keywords: Pediatrics; All-in-One; Wireless; Pateint remote monitoring; SpO2; Pulse oximeter; Skin Colour; VT-Patch

STUDY DESIGN:
Intervention Model Description: Monitoring of vital signs with VT-Patch and standard of care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monitored children (Experimental): PICU Children that will be monitored with the device
  Interventions: Device: Monitoring with VT-Patch (Connected device manufactured by VitalTracer)

INTERVENTIONS:
Device: Monitoring with VT-Patch (Connected device manufactured by VitalTracer) — Patients will be monitored for 8 consecutive hours and vital signs will be recorded with VT-Patch and with the standard of care

SUMMARY:
Small connected devices monitoring vital signs do not exist in children although they could be very useful to monitor patients once they have left the pediatric intensive care unit (PICU) in order to early identify patients at risk of PICU readmission.

The main objective of this study is to assess the accuracy of a connected thoracic patch (VT-Patch) for the continuous monitoring of vital signs in PICU patients.

This monitoring device will be used to monitor children in PICU for 8 hours and results will be compared to the standard of care in the unit which is the Philips monitoring system.

The investigators will assess the device's accuracy for the monitoring of 4 vital signs (SpO2, heart rate, respiratory rate and temperature) and perform exploratory assessment of three additional parameters (EKG, blood pressure and movement capture). The skin colour of each participant will be categorized based on Fitzpatrick scale and non-invasive spectroscopic method.

DETAILED DESCRIPTION:
Introduction:

Patients readmission to PICU is a major point of concern for physician because, although being a rare event, it has been strongly associated to more morbidity and death. Patients monitoring once they have left the PICU is drastically modified and small connected devices could be an option to early identify patients at risk of PICU readmission. Such devices have been manufactured for the monitoring of adults but they do not exist for children.

Besides, studies have recently shown that devices that use optical sensors may be less accurate in individuals with dark skin pigmentation since dark skin tones impose a limitation on optical biometric sensing. The wearable and medical device industry has not sufficiently addressed this issue yet. This is one of the main challenges that need to be addressed in this area to make sure the connected devices using this technology will work with all different skin colours including very dark skin.

Main objective:

Assess the accuracy of VT-Patch to measure oxygen saturation (SpO2) in children with diverse skin colour.

Secondary objectives:

Assess the accuracy of VT-Patch monitoring for 3 additional physiologic parameters (heart rate (HR), respiratory rate (RR) and temperature). Exploratory assessment of blood pressure (BP) monitoring, ECG signal and movement capture. The effect of the skin colour on the vital signs measurements will be investigated as well.

Design:

Prospective validation study of VT-Patch device for the monitoring of 4 physiologic parameters and exploratory assessment of three additional parameters.

Methods:

The study will be performed in two successive phases:

* Run-in phase: testing the device on 5 children to assess the feasibility of the protocol.
* Main study: validation phase of the device on 2 children per age group per skin phototype (based on Monk scale) to assess its accuracy. The patients of the run-in phase will be included in the main study if no modification of the protocol is required.

  4 physiologic parameters (HR, SpO2, RR, temperature and BP) and ECG will be prospectively recorded during 8 hours with VT-Patch and the regular monitoring system implemented in the unit High-resolution database that will be the Gold standard for evaluation.

Participating center: 1 center (St. Justine's Hospital).

Perspectives: This validation step of the collected data is necessary to validate that VT-Patch is suitable for pediatric patient monitoring of all skin colors.

ELIGIBILITY:
Inclusion Criteria:

* Children (0 to 18 years old) admitted in St. Justine's Hospital's PICU.
* PICU monitoring for the next 24 hours

Exclusion Criteria:

* Recent cardiac or thoracic surgery
* Thoracic skin lesion that contraindicates the VT-Patch
* No parental consent
* Intermittent presence of one study observer in the patient room is considered inappropriate by the physician or the nurse in charge because of the child's medical condition

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
SpO2 | 8 hours
  Percentage of the difference between the absolute value of SpO2 recorded by VT-Patch and the one recorded using standard of care

SECONDARY OUTCOMES:
Heart rate | 8 hours
  Percentage of the difference between the absolute value of heart rate recorded by VT-Patch and the one recorded using the standard of care
Respiratory rate | 8 hours
  Percentage of the difference between the absolute value of respiratory rate recorded by VT-Patch and the one recorded using standard of care
Temperature | 8hours
  Percentage of the difference between the absolute value of temperature recorded by VT-Patch and the one recorded using standard of care

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Jouvet, MD, PhD, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte Justin Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No